CLINICAL TRIAL: NCT04790500
Title: Effects Of Muscle Energy Technique Versus Mobilization On Pain And Disability In Post-Partum Females With Sacroiliac Joint Dysfunction.
Brief Title: Effects Of Muscle Energy Technique Versus Mobilization
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC/00846 Nusrat Javed
Record Dates: First submitted 2021-03-07; First posted 2021-03-10 (Actual); Last update posted 2021-09-23 (Actual); Status verified 2021-09

CONDITIONS: Sacroiliac Joint Dysfunction
Keywords: Mobilization; Muscle energy technique; Postpartum; Sacroiliac joint pain

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Active Comparator): mobilization technique
  Interventions: Other: mobilization technique
- Group B (Experimental): muscle energy technique
  Interventions: Other: muscle energy technique

INTERVENTIONS:
Other: mobilization technique — Mobilization of sacroiliac joint which will increase the range of motion and reduction in pain and improvement in functional limitation.
  Arms: Group A
Other: muscle energy technique — Muscle energy technique it is known as active muscular relaxation technique. It helps in lengthening the shorten muscle and increasing range of restricted muscles
  Arms: Group B

SUMMARY:
The aim is to describe the severity of pain in postpartum female and management of sacroiliac joint pain and disability and define the effects of manual therapy on sacroiliac joint dysfunction and pain

DETAILED DESCRIPTION:
The aim is to describe the severity of pain in postpartum female and management of sacroiliac joint pain and disability and define the effects of manual therapy on sacroiliac joint dysfunction and pain in postpartum females and to check whether the amount of gaining range of movement is similar among postpartum female undergoing with mobilization therapy and with muscle energy technique.

ELIGIBILITY:
Inclusion Criteria:

* 20-40 year having unilateral back pain around or on sacral sulcus,
* Positive posterior pain provocation test for Sacroiliac joint dysfunction,
* Low back pain within six weeks of delivery
* Pain while sitting down, lying on the ipsilateral side of pain, or climbing stairs.
* Local tenderness of the posterior aspect of the sacroiliac joint
* Pain is usually localized over the buttock.
* Sharp, stabbing, and/or shooting pain which extends down the posterior thigh usually not past the knee.
* C-section

Exclusion Criteria:

* Neurological deficit
* Spinal tumors
* Scoliosis,
* Underwent spinal surgery and prolapsed
* Intervertebral disc with or without radiculopathy

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2020-10-14 (Actual); Primary Completion 2021-08-20 (Actual); Study Completion 2021-08-20 (Actual)

PRIMARY OUTCOMES:
Numeric pain rating scale | 4th week
  o The 11-point (numeric pain rating scale) NPRS will use to capture the patient's level of pain. The scale is anchored on the left with the phrase ''no pain'' and on the right with the phrase ''worst imaginable pain.'' Patients rate their current level of pain and their worst and least amount of pain in the last 24 hours. The average of the 3 ratings or any single rating may be used to represent the patient's level of pain. Numeric pain scales have been shown to be reliable and valid. The reliability of numeric pain rating scale is 0.74
Modified Oswestry disability index | 4th week
  It is a self-report questionnaire of a patient's perceived disability based on 10 areas of pain and daily activities (pain intensity, personal hygiene, lifting, walking, sitting, standing, sleeping, sexual activity, social activity and travelling). Each section is scored on a6-point scale (0-5), with 0 representing no limitation and 5 representing maximal limitation. The subscales combined add up to a total maximal score of 50. The score is then doubled and interpreted as a percentage of the patient-perceived disability (the higher the score, the greater the disability). In cases where patients did not answer all the 10 sections, the sum score of the answered sections were divided by the number of completed sections. The reliability of modified oswestry disability index is 0.88.

CONTACTS AND LOCATIONS:
Overall Officials: Anam Aftab, Phd*, Principal Investigator — Riphah college of rehabilitation and allied health sciences - Rawalpindi
Locations (1):
- Pakistan railway hospital, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No